CLINICAL TRIAL: NCT00993226
Title: An International, Randomised, Double Blinded, Multi-centre, Active- and Placebo-controlled Dose Response Trial to Evaluate the Efficacy and Safety of SABER-Bupivacaine for Postoperative Pain Control in Patients Undergoing Primary, Elective, Open, Abdominal Hysterectomy
Brief Title: An International Trial to Evaluate the Efficacy and Safety of SABER®-Bupivacaine for Postoperative Pain Control in Patients Undergoing Hysterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: Nycomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BU-001-IM
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Local anaesthesia; Postoperative pain after open abdominal hysterectomy surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- SABER-Bupivacaine Treatment 1a (Experimental): double-blind
  Interventions: Drug: SABER-Bupivacaine Treatment 1a
- Placebo SABER-Bupivacaine Treatment 1b (Placebo Comparator): double-blind
  Interventions: Drug: Placebo SABER-Bupivacaine Treatment 1b
- Bupivacaine HCl Treatment 1c (Active Comparator): double-blind
  Interventions: Drug: Bupivacaine HCl Treatment 1c
- SABER-Bupivacaine Treatment 2a (Experimental): double-blind
  Interventions: Drug: SABER-Bupivacaine Treatment 2a
- Placebo SABER-Bupivacaine Treatment 2b (Placebo Comparator): double-blind
  Interventions: Drug: Placebo SABER-Bupivacaine Treatment 2b
- Bupivacaine HCl Treatment 2c (Active Comparator): double-blind
  Interventions: Drug: Bupivacaine HCl Treatment 2c

INTERVENTIONS:
Drug: SABER-Bupivacaine Treatment 1a — 5.0 ml
  Arms: SABER-Bupivacaine Treatment 1a
Drug: Placebo SABER-Bupivacaine Treatment 1b — 5.0 ml
  Other Names: POSIMIR® bupivacaine solution
  Arms: Placebo SABER-Bupivacaine Treatment 1b
Drug: Bupivacaine HCl Treatment 1c — 40 ml
  Arms: Bupivacaine HCl Treatment 1c
Drug: SABER-Bupivacaine Treatment 2a — 7.5 ml
  Arms: SABER-Bupivacaine Treatment 2a
Drug: Placebo SABER-Bupivacaine Treatment 2b — 7.5 ml
  Arms: Placebo SABER-Bupivacaine Treatment 2b
Drug: Bupivacaine HCl Treatment 2c — 40 ml
  Arms: Bupivacaine HCl Treatment 2c

SUMMARY:
The objective is to identify the optimal dose of SABER-Bupivacaine for postoperative pain control in patients undergoing hysterectomy on the basis of pharmacokinetics, efficacy and safety evaluations. The study duration consists of a screening period up to 14 days and a treatment period 14 days with a long term follow up visit at 6 months. The study will provide further data on the efficacy and safety of the product.

ELIGIBILITY:
Inclusion Criteria:

* A planned elective, abdominal hysterectomy
* Patients suitable for general anaesthesia

Exclusion Criteria:

* Known clinically significant hepatic, gastrointestinal, renal, haematological, urologic, neurological, respiratory, endocrine or cardiovascular system abnormalities
* Known serious uncontrolled illness: cancer, psychiatric or metabolic disturbances. History of cured localised malignancies is allowed (i.e. basal or squamous cell skin carcinoma, breast carcinoma or cervical carcinoma)
* Abnormal ECG
* Prolonged QT syndrome
* Current or regular use of analgesic medication for other indication(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquarters
Locations (14):
- Nycomed, Paris, France
- Germany (2):
  - Nycomed, Bayreuth
  - Nycomed, Dresden
- Hungary (8):
  - Nycomed, Békéscsaba
  - Nycomed, Budapest
  - Nycomed, Debrecen
  - Nycomed, Győr
  - Nycomed, Nyíregyháza
  - Nycomed, Székesfehérvár
  - Nycomed, Szolnok
  - Nycomed, Tatabánya
- Nycomed, Riga, Latvia
- Nycomed, Stockholm, Sweden
- Nycomed, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- SABER-Bupivacaine; SABER-placebo: 5 mL, single dose instilled into surgical incision
- Bupivacaine HCl: 0.25% 40 mL, single dose infiltrated peri-incisionally
Period: Overall Study
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Started | 61 | 27 | 27
Completed | 60 | 26 | 27
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl | Total
Number analyzed (Participants) | 61 | 27 | 27 | 115
Age, Continuous [Mean (Full Range); unit: years] | 46.7 [29 to 66] | 44.3 [37 to 53] | 45.1 [35 to 55] | 45.8 [29 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 27 | 27 | 115
  Male | 0 | 0 | 0 | 0
BMI [Mean (Full Range); unit: kg/m^2] | 26.1 [19.0 to 33.2] | 26.2 [19.4 to 34.1] | 27.0 [18.3 to 35.0] | 26.4 [18.3 to 35.0]

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity (PI)
Description: Pain intensity (PI) on movement AUC over the period 1 to 72 hours post-surgery. Subjects assessed their pain intensity using an 11-point Pain Intensity Numeric Rating Scale (PI-NRS) with NRS scores ranging from 0 (no pain) to 10 (worst pain possible). The AUC is computed for each patient using the standard trapezoidal rule and normalised by dividing by the time interval over which it is computed. This normalisation converts the AUC to the natural pain scale (NRS 0-10) to allow for better translation of the clinical treatment effect magnitude.
Time Frame: 1 to 72 hours post-surgery
Population: ITT population (patients with data available)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Number analyzed (Participants) | 60 | 27 | 27
score on a scale | 4.15 (1.74) | 4.46 (1.48) | 4.27 (1.69)
Statistical Analysis 1: Comparison: SABER-Bupivacaine vs SABER-placebo; Exploratory comparison between SABER-Bupivacaine and Bupivacaine HCl not analyzed inferentially; Test type: Superiority; p = 0.467, t-test in ANOVA model; LS Mean Difference = -0.21, 95% CI 2-sided [-0.79 to 0.36], Standard Deviation 0.29

2. Primary Outcome: Supplemental Opioid Use
Description: Cumulative IV morphine-equivalent dose of opioid rescue medication
Time Frame: 0-3 days after surgery
Population: ITT population (patients with data available)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Number analyzed (Participants) | 61 | 27 | 27
mg | 22.8 (24.3) | 26.3 (25.7) | 23.9 (25.9)
Statistical Analysis 1: Comparison: SABER-Bupivacaine vs SABER-placebo; Exploratory comparison between SABER-Bupivacaine and Bupivacaine HCl not analyzed inferentially; Test type: Superiority; p = 0.331, t-test in ANOVA model; LS Mean Difference = -2.51, 95% CI 2-sided [-7.59 to 2.58], Standard Deviation 2.57

3. Secondary Outcome: Time to First Opioid Rescue Medication Usage
Time Frame: 0-14 days after surgery
Population: ITT population (patients with data available)
Measure: Median (Standard Deviation); unit: hours
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Number analyzed (Participants) | 61 | 27 | 27
hours | 7.71 (45.79) | 1.53 (1.56) | 87.77 (1.11)

4. Secondary Outcome: Opioid Related Side Effects
Description: Opioid-related side effects were recorded 0-7 days after surgery. The Opioid-Related Symptom Distress Scale (OR-SDS) is a composite score computed from a questionnaire containing frequent opioid-related symptoms (Fatigue, Drowsiness, Inability to concentrate, Nausea, Dizziness, Constipation, Itching, Difficulty with urination, Confusion, Retching/vomiting). For each symptom, patients assigned integer scores to assess severity (none=0 to very severe=4), bothersomeness (none=0 to very much=5), and frequency (none=0 to almost constantly=4); patients reported number of Retching/vomiting episodes (none=0, 1-2 episodes=1, 3-4 episodes=2, 5-6 episodes=3, >6 episodes=4).
  On each day (Day 0-7), the score for each symptom was the mean of the three component scores, and the OR-SDS score was the overall mean of the 10 symptom scores, (values from 0 to 4; larger outcomes are worse). The mean of the daily OR-SDS score from Day 0 to 7 gave the overall OR-SDS Score.
Time Frame: 0-7 days after surgery
Population: ITT population (patients with data available)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
Number analyzed (Participants) | 53 | 25 | 23
score on a scale | 0.28 (0.28) | 0.34 (0.31) | 0.27 (0.24)

ADVERSE EVENTS:
Arm/Group | SABER-Bupivacaine | SABER-placebo | Bupivacaine HCl
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 7/60 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 48/60 | 17/27 | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SABER-Bupivacaine (N=60) | SABER-placebo (N=27) | Bupivacaine HCl (N=27)
ECG abnormal (Investigations) | 2 | 0 | 0
ECG QT prolonged (Investigations) | 1 | 0 | 0
Haematoma infection (Infections and infestations) | 2 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SABER-Bupivacaine (N=60) | SABER-placebo (N=27) | Bupivacaine HCl (N=27)
Post procedural contusion (Injury, poisoning and procedural complications) | 36 | 9 | 0
Anaemia (Blood and lymphatic system disorders) | 10 | 4 | 3
Vomiting (Gastrointestinal disorders) | 9 | 8 | 4
Dizziness (Nervous system disorders) | 9 | 3 | 4
Pyrexia (General disorders) | 7 | 3 | 7
CRP increased (Investigations) | 7 | 0 | 1
Somnolence (Nervous system disorders) | 5 | 0 | 2
Blood potassium decreased (Investigations) | 4 | 1 | 0
Hypertension (Vascular disorders) | 4 | 1 | 2
Incision site haematoma (Injury, poisoning and procedural complications) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes